CLINICAL TRIAL: NCT04896073
Title: A Phase II Trial of the Superenhancer Inhibitor Minnelide in Advanced Refractory Adenosquamous Carcinoma of the Pancreas (ASCP)
Brief Title: Superenhancer Inhibitor Minnelide in Advanced Refractory Adenosquamous Carcinoma of the Pancreas (ASCP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anish Thomas, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000254; 000254-C
Record Dates: First submitted 2021-05-20; First posted 2021-05-21 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Adenosquamous Carcinoma of the Pancreas
Keywords: Pancreatic Ductal Adenocarcinoma; epigenetic changes; MYC; triptolide; HSP70
MeSH Terms: interventions — 14-O-phosphonooxymethyltriptolide disodium salt; Electrocardiography; Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP) (Experimental): Minnelide 2mg Days 1-21 of 28-day cycle (x12)
  Interventions: Drug: Minnelide; Diagnostic Test: ECG; Diagnostic Test: CT/MRI; Procedure: Tumor Biopsy

INTERVENTIONS:
Drug: Minnelide — Administered orally (2 mg) once daily for 21 days of 28-day cycles for 12 cycles.
  Other Names: 14-O-phosphonooxymethyltriptolide-disodium-salt and Minnelide-001
Diagnostic Test: ECG — Screening and end of treatment visit.
  Other Names: Electrocardiogram
Diagnostic Test: CT/MRI — Screening. Subsequent cycles Day 1 (≤3days) and Day 15 (±2 days) (every other cycle). End of treatment visit.
  Other Names: Computed tomography/Magnetic resonance imaging
Procedure: Tumor Biopsy — Optional. Baseline Cycle 1, Day 1 and Cycle 1, Day 15. End of treatment visit or progressive disease.
  Other Names: Tumor Bx

SUMMARY:
Background:

Pancreatic cancer is one of the most lethal types of cancer. American Society for Clinical Pathology (ASCP) is a highly aggressive type of pancreatic cancer. It is very rare. Researchers want to see if a drug called Minnelide can be used to treat ASCP.

Objective:

To see if Minnelide is an effective treatment for ASCP.

Eligibility:

Adults ages 18 and older with ASCP whose cancer did not respond to previous treatments.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine samples

Evaluation of ability to do daily activities

Electrocardiogram to test heart function

Body and/or brain scans. For these, participants will lie in a machine that takes pictures of the body. They may have a contrast agent injected into a vein.

Tumor sample. If one is not available, participants will have a tumor biopsy. The biopsy will be taken with a small needle put through the skin into the tumor.

Treatment will be given in 28-day cycles, for up to 12 cycles. There is a 7-day resting period between cycles. Participants will take Minnelide by mouth every day for 21 days of each cycle. They will keep a medicine diary.

Participants will have at least 1 study visit every cycle. They will review their medicine diary. They will repeat some screening tests.

Participants may have optional tumor biopsies. Some participants may need to take birth control during the study and for up to 6 months after treatment.

Participants will have an end-of-treatment visit 4 weeks after they stop taking the study drug. They will repeat some screening tests.

DETAILED DESCRIPTION:
Background:

* Adenosquamous carcinoma of the pancreas (ASCP) is a highly aggressive variant of pancreatic ductal adenocarcinoma (PDA), the most common type of pancreas cancer.
* ASCP is estimated to account for 0.5-4% of the 55,000 people who are diagnosed with pancreatic cancer in the United States (U.S.) each year, making it a very rare tumor type.
* No prospective clinical trials specific to ASCP have ever been performed.
* Preclinical data in ASCP models indicate that an activated superenhancer network drives epigenetic changes which cause the prognostically unfavorable squamous differentiation.
* Genomic analysis of ASCP tumors identifies frequent amplification of MYC.
* Minnelide is a small molecule anti-superenhancer drug that inhibits MYC.
* The recommended dose of Minnelide has previously been established through clinical testing for other indications.

Primary Objective:

-To determine the single agent antitumor activity (disease control rate) of the anti-superenhancer agent Minnelide in participants with advanced, previously treated ASCP

Eligibility:

* Age >= 18 years
* Histologically confirmed ASCP or high suspicion for ASCP based on histologic analysis for squamous markers
* Participants with metastatic or locally advanced unresectable disease and progression on at least 1 prior treatment regimen

Design:

* This is a phase II single cohort clinical trial with one arm.
* The number of evaluable participants needed for the primary endpoint is 25; maximum accrual set at 55 participants (accounting for screen failures and inevaluable participants).
* initial participants will receive Minnelide at 2 mg/day by mouth (PO) on Days 1-21 of a 28-day cycle.
* Later participants will receive a higher dose of 2.5 mg/day PO on the same schedule.
* Treatment will be continued for up to 12 cycles (1 year) in the absence of disease progression or unacceptable toxicity.
* Treatment response will be assessed by imaging every 2 cycles (8 weeks).
* Optional tumor biopsies will be requested mid-cycle 1 and at time of progression.
* A disease control rate of >= 40% in this highly refractory population would constitute a positive study. Up to 12 participants will be treated initially. If 3 of the 12 participants have a response, then up to 13 additional participants will be entered to determine the true response rate.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histological or cytological diagnosis of adenosquamous carcinoma of the pancreas (ASCP) or high suspicion for ASCP as confirmed by National Institutes of Health (NIH) Laboratory of Pathology. ASCP will be defined as >=30% malignant squamous component in background of typical pancreatic ductal adenocarcinoma (PDA). If malignant squamous component is identified in the sample, but the pathologist is unable to determine whether it is >= 30%, then the participant will be considered to have high suspicion for ASCP.

Note: To meet this criterion, participant must be able to submit a suitable archival tumor specimen (primary or metastatic site) for review or currently have tumor in a location deemed low risk for core biopsy so that suitable tissue can be acquired for confirmation of diagnosis. Note that cytopathology specimens are not considered suitable for definitive diagnosis of ASCP but can be used to determine high suspicion for ASCP.

* Participants with metastatic, recurrent or locally advanced unresectable disease and progression or intolerance to at least 1 prior systemic treatment regimen in the advanced disease setting.
* Disease measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Progressive disease as evidenced by increasing tumor size on radiologic assessment, increasing serum tumor marker (on last 2 measurements taken at least 1 week apart), increasing ascites, and/or worsening tumor-related symptoms such as weight loss, pain, gastrointestinal (GI) upset.
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%).
* Be willing and able to provide written informed consent for the trial.
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count (ANC) >= 1,500/microL
  * platelets >= 100,000/microL
  * hemoglobin >= 9.0 g/dL or >= 5.6 mmol/La*
  * Creatinine <= 1.5 x ULN

OR

measured or calculated *bcreatinine clearance (Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl) >= 45 mL/min for participant with creatinine levels >1.5 x institutional upper limit of normal (ULN)

* total bilirubin <= 1.5 x ULN OR direct bilirubin <= ULN for participants with total bilirubin levels >1.5 x ULN
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) <= 2.5 x ULN (<= 5 x ULN for participants with liver metastases)
* International normalized ratio (INR) OR

  * prothrombin time (PT)
  * activated partial thromboplastin time (aPTT):

<= 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT) = alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT) = aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR = glomerular filtration rate; ULN=upper limit of normal.

*a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC)

transfusion within last 2 weeks.

*b Creatinine clearance (CrCl) should be calculated per institutional standard.

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

-The effects of Minnelide on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months (women) and 3 months (men) after the last dose of trial treatment. Male participants must also refrain from donating sperm during this period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Has uncontrolled vomiting or medical condition which inhibits oral ingestion or digestion because the study treatment is administered orally.
* Pregnant and/or women who are breast feeding are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Minnelide.
* Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent/therapy or used an investigational device within 3 weeks of the first planned treatment on this study.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1/Day 1
* Requires use of ondansetron or another prohibited medication. Note that other 5-hydroxytryptamine 3 (5-HT3) inhibitors are NOT prohibited.
* Has received major surgery within the last 4 weeks, minor endoscopic procedure such as biliary stenting within the last 2 weeks, or percutaneous procedure such as hepatic biopsy or celiac plexus block within 24 hours of planned treatment start date. Note: participant must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

Participants with previously treated brain metastases may participate if:

a) follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression at >= 4 weeks since treatment, AND b) participant has stability of baseline neurologic symptoms without receiving immunosuppressive-doses of systemic corticosteroid (physiologic replacement doses are permitted) x7 days or increases in other supportive medications that treat neurologic symptoms such as antiepileptics x14 days. Participants with carcinomatous meningitis are excluded regardless of clinical stability.

* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant s participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has known uncontrolled or poorly controlled human immunodeficiency virus (HIV) infection. HIV is considered uncontrolled or poorly controlled if an HIV-infected individual is not taking highly active anti-retroviral therapy or has a detectable viral load within the previous 6 months.
* Has active hepatitis B virus (HBV) or hepatitis C virus (HCV) or is currently under treatment for HBV or HCV. Active HBV or HCV does not include previously cleared HBV or HCV or successfully cured HBV or HCV through treatment
* Has received a live vaccine within 30 days of planned start of trial therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist (Registered Trademark)) are live attenuated vaccines and are not allowed.

-History of allergic reactions attributed to compounds of similar chemical or biologic composition to Minnelide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data is available once genomic data is uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data is made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Skorupan N, Ahmad MI, Steinberg SM, Trepel JB, Cridebring D, Han H, Von Hoff DD, Alewine C. A phase II trial of the super-enhancer inhibitor Minnelide in advanced refractory adenosquamous carcinoma of the pancreas. Future Oncol. 2022 Jun;18(20):2475-2481. doi: 10.2217/fon-2021-1609. Epub 2022 May 10. PMID 35535581
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000254-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled, Not Assigned to a Cohort and Not Treated: Participants were enrolled, not assigned to a Cohort and not treated.
Period: Overall Study
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP) | Enrolled, Not Assigned to a Cohort and Not Treated
Started | 12 | 4
Completed | 12 | 0
Not Completed | 0 | 4
Not completed — Screen failure | 0 | 2
Not completed — Participant declined to participate (before treatment started) | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for participants enrolled, not assigned to a Cohort and not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP) | Enrolled, Not Assigned to a Cohort and Not Treated | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.58 (11.44) | 59.75 (12.66) | 65.63 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 4 | 14
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 2 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Evaluable Participants Who Experience Clinical Benefit (Disease Control Rate = Complete Response (CR)+Partial Response (PR)+Stable Disease x16 Weeks) Reported Along With a 95% Confidence Interval
Description: To determine the single agent antitumor activity (disease control rate = CR + PR + stable disease x16 weeks) of the anti-superenhancer agent Minnelide in participants with advanced, previously treated adenosquamous carcinoma of the pancreas (ASCP) using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of diameters while on study. Progressive Disease is least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: 16 weeks
Population: 12/16 participants were analyzed because 2 were screen failures and 2 declined to participate before treatment started.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
Number analyzed (Participants) | 12
Proportion of participants
  Complete Response | 0 [0 to 0]
  Partial Response | 0 [0 to 0]
  Stable Disease | .0083 [0.002 to 0.385]

2. Secondary Outcome: Number of Participants Who Experience a Non-serious Grade 2 or Higher Toxicity, by Grade and Type of Toxicity Assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Description: Non-serious adverse events of Minnelide were assessed by the Common Terminology Criteria for Adverse Events (CTCAE). A non-serious adverse event is any untoward medical occurrence. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse events.
Time Frame: Non-serious adverse events related to Minnelide that occur from start of treatment to 30 days after last treatment
Measure: Count of Participants; unit: Participants
Groups:
- Grade 2; Grade 3; Grade 4; Grade 5: Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
  Minnelide 2mg Days 1-21 of 28-day cycle (x12)
  Minnelide: Administered orally (2 mg) once daily for 21 days of 28-day cycles for 12 cycles.
Arm/Group | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Abdominal pain | 2 | 1 | 0 | 0
  Anemia | 6 | 5 | 1 | 0
  Anorexia | 3 | 2 | 0 | 0
  Ascites | 1 | 1 | 0 | 0
  Bloating | 1 | 0 | 0 | 0
  Blood bilirubin increased | 1 | 1 | 0 | 0
  Chills | 1 | 0 | 0 | 0
  Creatinine increased | 1 | 0 | 0 | 0
  Dehydration | 1 | 0 | 0 | 0
  Diarrhea | 2 | 0 | 0 | 0
  Encephalopathy | 1 | 0 | 1 | 0
  Enterocolitis infectious | 0 | 1 | 0 | 0
  Eye disorders - Other, specify - corneal abrasion of the right eye | 1 | 0 | 0 | 0
  Fall | 3 | 0 | 0 | 0
  Fatigue | 3 | 1 | 0 | 0
  Hiccups | 1 | 0 | 0 | 0
  Hypercalcemia | 1 | 1 | 0 | 0
  Hypoalbuminemia | 4 | 0 | 0 | 0
  Hypoglycemia | 1 | 0 | 0 | 0
  Hypokalemia | 1 | 0 | 0 | 0
  Hyponatremia | 0 | 1 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0 | 0
  Hypotension | 0 | 1 | 0 | 0
  Malaise | 2 | 0 | 0 | 0
  Nausea | 5 | 3 | 0 | 0
  Neutrophil count decreased | 2 | 2 | 1 | 0
  Oropharyngeal pain | 1 | 0 | 0 | 0
  Pain | 1 | 0 | 0 | 0
  Platelet count decreased | 3 | 2 | 3 | 0
  Pleural effusion | 1 | 0 | 0 | 0
  Presyncope | 1 | 0 | 0 | 0
  Syncope | 0 | 1 | 0 | 0
  Upper gastrointestinal hemorrhage | 0 | 1 | 0 | 0
  Upper respiratory infection | 1 | 0 | 0 | 0
  Vomiting | 2 | 3 | 0 | 0
  White blood cell decreased | 0 | 2 | 2 | 0

3. Secondary Outcome: Number of Participants Who Experience a Serious Grade 2 or Higher Toxicity, by Grade and Type of Toxicity Assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Description: Serious adverse events of Minnelite were assessed by the Common Terminology Criteria for Adverse Events (CTCAE). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse events.
Time Frame: Serious adverse events related to Minnelide that occur from start of treatment to 30 days after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Abdominal pain | 0 | 1 | 0 | 0
  Anemia | 0 | 1 | 0 | 0
  Dehydration | 0 | 1 | 0 | 0
  Dyspnea | 1 | 0 | 0 | 0
  Encephalopathy | 0 | 0 | 0 | 1
  Enterocolitis | 0 | 1 | 0 | 0
  Nausea | 0 | 1 | 0 | 0
  Nervous system disorders - Other specify - balance difficulty | 1 | 0 | 0 | 0
  Stroke | 0 | 0 | 0 | 1
  Thromboembolic event | 0 | 1 | 0 | 0
  Upper gastrointestinal hemorrhage | 0 | 1 | 0 | 0
  Urinary tract infection | 0 | 1 | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. PFS will be determined using the Kaplan-Meier method and reported along with a 95% confidence interval for the median. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Progressive Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: start of treatment to time of progression or death, a median of 1.76 months
Population: 12/16 participants were analyzed because 2 were screen failures and 2 declined to participate before treatment started.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
Number analyzed (Participants) | 12
Months | 1.76 [0.90 to 2.62]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the length of time from the start of treatment until death. OS will be determined by using the Kaplan-Meier method and reported along with a 95% confidence interval for the median.
Time Frame: time from the start of treatment until death, a median of 4.91 months
Population: 12/16 participants were analyzed because 2 were screen failures and 2 declined to participate before treatment started.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
Number analyzed (Participants) | 12
Months | 4.91 [1.96 to 7.85]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) will be calculated as the percentage of participants with Complete Response (CR) or Partial Response (PR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST)1.1 criteria. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From start of treatment until radiological progression response or off study; the median is approximately 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
Number analyzed (Participants) | 12
percentage of participants
  Complete Response | 0
  Partial Response | 0

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events were monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered
Population: 12/16 participants were analyzed because 2 were screen failures and 2 declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered
Description: 12/16 participants were analyzed because 2 were screen failures and 2 declined to participate before treatment started.
Arm/Group | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP)
All-Cause Mortality (participants affected / at risk) | 11/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP) (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, specify: balance difficulty (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1, Minnelide in Advanced Adenosquamous Carcinoma of the Pancreas (ASCP) (N=12)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (20)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Ascites (Gastrointestinal disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2)
Chills (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (2)
Enterocolitis infectious (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, specify: corneal abrasion of the right eye (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 2 (3)
Generalized edema (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (11)
Neutrophil count decreased (Investigations) | 3 (6)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Platelet count decreased (Investigations) | 5 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9)
White blood cell decreased (Investigations) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-07-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT04896073/Prot_SAP_000.pdf
  • Informed Consent Form: Redacted Cohort Affected Patient Screening Consent (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT04896073/ICF_001.pdf
  • Informed Consent Form: Redacted Cohort Affected Patient Standard Consent (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT04896073/ICF_002.pdf